CLINICAL TRIAL: NCT01114737
Title: A Double-blind, Placebo-controlled, Randomized Study to Evaluate the Safety and Therapeutic Effects of Sapropterin Dihydrochloride on Neuropsychiatric Symptoms in Subjects With Phenylketonuria
Brief Title: Safety and Therapeutic Effects of Sapropterin Dihydrochloride on Neuropsychiatric Symptoms in Phenylketonuria (PKU) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PKU-016; PKU Ascend (Other: BioMarin Pharmaceutical)
Record Dates: First submitted 2010-04-27; First posted 2010-05-03 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; PKU; Kuvan; Sapropterin dihydrochloride; Neuropsychiatric disorder; ADHD
MeSH Terms: conditions — Phenylketonurias; Attention Deficit Disorder with Hyperactivity | interventions — sapropterin; phenoptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sapropterin dihydrochloride (Experimental)
  Interventions: Drug: Sapropterin dihydrochloride
- Tablet without active ingredient (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sapropterin dihydrochloride — A dose of 20 mg/kg/day will be administered. Route of administration is oral (intact).
  Other Names: Kuvan; Phenoptin; BH4; 6R BH4
  Arms: Sapropterin dihydrochloride
Drug: Placebo — Placebo (tablet without active ingredient) is dosed once/day for the first 13 weeks of the study.
  Arms: Tablet without active ingredient

SUMMARY:
This double-blind, placebo-controlled, randomized study is designed to evaluate the safety and therapeutic effects of sapropterin dihydrochloride on neuropsychiatric symptoms in subjects with PKU.

DETAILED DESCRIPTION:
Phenylketonuria (PKU) results from deficient phenylalanine hydroxylase (PAH) activity and leads to toxic phenylalanine (Phe) accumulation in patients with PKU causing mental retardation, microcephaly, delayed speech, seizures, psychiatric symptoms and behavioral abnormalities. Although for most PKU patients early initiation of dietary treatment prevents severe complications, discontinuation of dietary restrictions at an early age is associated with poor cognitive development and neuropsychiatric disorders are present even in early-treated and well controlled PKU patients.

This study, PKU-016, will be conducted in PKU patients to evaluate the therapeutic effects of sapropterin dihydrochloride on the symptoms of attention deficit hyperactivity disorder (ADHD), depression, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 8 years of age
* Confirmed diagnosis of PKU
* Willing to continue current diet (typical diet for the 3 months prior to study entry) unchanged while participating in the study
* Willing and able to provide written, signed informed consent or in the case of subjects under the age of 18, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study and for at least 30 days following the last dose of sapropterin dihydrochloride
* Females of childbearing potential must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to screening, or have had total hysterectomy.
* Willing and able to comply with all study procedure

Exclusion Criteria:

* Has known hypersensitivity to sapropterin dihydrochloride or its excipients
* Subject breastfeeding at screening or planning to become pregnant (subject or partner) at any time during the study
* Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to the completion of all scheduled study assessments
* Received sapropterin dihydrochloride within 16 weeks of randomization
* Have initiated or adjusted medication for treatment of ADHD, depression, or anxiety ≤ 8 weeks prior to randomization
* Taking medication known to inhibit folate synthesis (eg, methotrexate)
* Any condition requiring treatment with levodopa or any PDE-5 inhibitor
* Concurrent disease or condition that would interfere with study participation, compliance or safety as determined by the Investigator
* Any condition that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suyash Prasad, MD, Study Director — BioMarin Pharmaceutical
Locations (36):
- United States (26):
  - La Jolla, California
  - Los Angeles, California
  - Palo Alto, California
  - San Francisco, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Albany, New York
  - Buffalo, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Grant ML, Jurecki ER, McCandless SE, Stahl SM, Bilder DA, Sanchez-Valle A, Dimmock D. Neuropsychiatric Function Improvement in Pediatric Patients with Phenylketonuria. J Pediatr. 2023 Sep;260:113526. doi: 10.1016/j.jpeds.2023.113526. Epub 2023 May 30. PMID 37263523

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: Placebo (tablet without active ingredient) is dosed once/day for the first 13 weeks of the study(double-blinded randomized treatment period); then treated with sapropterin dihydrochloride 20 mg/kg/day for an additional 13 weeks (open label treatment period).
- 6R-BH4 20 mg/kg/Day: Sapropterin dihydrochloride: A dose of 20 mg/kg/day will be administered. Route of administration is oral (intact). Patient will be treated for 26 weeks, the first 13 weeks were double-blinded randomized treatment period, the second 13 weeks open label treatment period
Period: Randomized Treatment Period
Arm/Group | Placebo | 6R-BH4 20 mg/kg/Day
Started | 108 | 98
Completed | 105 | 97
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Pregnancy | 1 | 0
Period: Open-Label Treatment Period
Arm/Group | Placebo | 6R-BH4 20 mg/kg/Day
Started | 105 (One subject did not receive a single dose of the study drug) | 97 (Two subjects did not receive a single dose of the study drug)
Completed | 100 | 95
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Difficult Personal Events | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 6R-BH4 20 mg/kg/Day | Total
Number analyzed (Participants) | 108 | 98 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (10.42) | 23.6 (12.69) | 23.1 (11.54)
Age, Customized [Number; unit: participants]
  <18 years | 43 | 43 | 86
  >=18 years | 65 | 55 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 41 | 95
  Male | 54 | 57 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 105 | 93 | 198
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 102 | 96 | 198
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 38 | 31 | 69
  United States | 70 | 67 | 137

OUTCOME MEASURES:

1. Primary Outcome: Change in Attention-Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS) / Adult ADHD Self-Report Scale (ASRS) Total Score From Baseline to Week 13
Description: Effects of 6R-BH4 on symptoms of ADHD in PKU subjects who had symptoms of ADHD at screening in the subjects that had a blood Phe level reduction after treatment with 6R-BH4.
  The total ADHD-RS score and the corrected total ARS score range from 0 to 54, with higher scores corresponding to worse severity of ADHD symptoms.
Time Frame: Baseline to Week 13
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Responders in Placebo Arm With ADHD Symptoms: Included all subjects in the Placebo arm who had a blood Phe level reduction ≥ 20% from Baseline within their first 4 weeks of sapropterin treatment with ADHD symptoms at Baseline
- Responders in 6R-BH4 20 mg/kg/Day Arm With ADHD Symptoms: Included all subjects in the 6R-BH4 20 mg/kg/day Arm who had a blood Phe level reduction ≥ 20% from Baseline within their first 4 weeks of sapropterin treatment with ADHD symptoms at Baseline
Arm/Group | Responders in Placebo Arm With ADHD Symptoms | Responders in 6R-BH4 20 mg/kg/Day Arm With ADHD Symptoms
Number analyzed (Participants) | 19 | 19
units on a scale | -4.9 [-8.9 to -0.9] | -9.1 [-13.5 to -4.7]
Statistical Analysis 1: Comparison: Responders in Placebo Arm With ADHD Symptoms vs Responders in 6R-BH4 20 mg/kg/Day Arm With ADHD Symptoms; Test type: Superiority or Other; p = 0.085, ANCOVA; Adjusted for baseline ADHD-RS/ASRS total score, age group, and ADHD medication; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-8.9 to 0.6], Standard Error of Mean 2.3

2. Secondary Outcome: Change in Hamilton Anxiety Rating Scale (HAM-A) Score From Baseline to Week 13
Description: Effects of 6R-BH4 on symptoms of anxiety in PKU subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  HAM-A Score is a total score ranging from 0 to 56 with higher scores corresponding to worse severity of anxiety symptoms. The HAM-A has 14 items, each measuring specific anxiety symptom clusters. Each item is given a 5-point-score as: 0, absent; 1, mild; 2, moderate; 3, severe; or 4, incapacitating.
Time Frame: Baseline to Week 13
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Responders in Placebo Arm: Included all subjects in the Placebo arm who had a blood Phe level reduction ≥ 20% from Baseline within their first 4 weeks of sapropterin treatment
- Responders in 6R-BH4 20 mg/kg/Day Arm: Included all subjects in the 6R-BH4 20 mg/kg/day Arm who had a blood Phe level reduction ≥ 20% from Baseline within their first 4 weeks of sapropterin treatment
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 61
units on a scale | -3.6 [-5.4 to -1.9] | -3.2 [-5.1 to -1.4]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.669, ANCOVA; Adjusted for baseline HAMA Anxiety Scale Total Score, age group, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.5 to 2.3], Standard Error of Mean 0.9

3. Secondary Outcome: Change in Hamilton Depression Rating Scale (HAM-D) Score From Baseline to Week 13
Description: Effects of 6R-BH4 on symptoms of depression in PKU subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  HAM-D Score is a total score ranging from 0 to 48 with higher scores corresponding to worse severity of depression. The HAM-D is a 17-item depression rating scale. Nine of the items are scored on a 5-point scale as: 0, absence of depressive symptom being measured; 1, doubt concerning the presence of the symptom; 2, mild symptoms; 3, moderate symptoms; or 4, severe symptoms. The remaining 8 items are scored on a 3-point scale as: 0, absence; 1, doubt on the presence of the symptom; or 2, clear presence of symptoms.
Time Frame: Baseline to Week 13
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 61
units on a scale | -2.5 [-3.9 to -1.1] | -2.1 [-3.6 to -0.6]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.588, ANCOVA; Adjusted for Baseline HAM-D Rating Scale Total Score, age group, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.1 to 1.9], Standard Error of Mean 0.8

4. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) From Baseline to Week 13
Description: Effects of 6R-BH4 on global function in PKU subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  CGI-S is a 7-point scale that requires the clinician to rate the severity of the subject's mental illness at the time of assessment, relative to clinician's past experience with subjects who have the same diagnosis. Considering total clinical experience, a subject is assessed on the severity of mental illness at the time of rating as: 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 6, severely ill; or 7, among the most extremely ill.
Time Frame: Baseline to Week 13
Population: Phe Responders
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 61
units on a scale | -0.5 [-0.8 to -0.2] | -0.6 [-0.9 to -0.3]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.531, ANCOVA; Adjusted for baseline CGI-Severity Response, age group, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.2

5. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF) Adult-Global Executive Composite (GEC) T Score From Baseline to Week 13
Description: Effects of 6R-BH4 on executive function in PKU subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  The scoring for the GEC T Score is complex and is achieved using proprietary software designed to generate scores based on raw data collected. Higher scores suggest a higher level of dysfunction.
Time Frame: Baseline to Week 13
Population: Phe Responders who are >=18 Years of Age
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 28 | 25
T score | -8.1 [-12.6 to -3.6] | -9.1 [-14.6 to -3.5]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.661, ANCOVA; Adjusted for Baseline BRIEF Adult-GEC T Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-5.5 to 3.6], Standard Error of Mean 2.2

6. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF) Parent-Global Executive Composite (GEC) T Score From Baseline to Week 13
Description: as for outcome 5
Time Frame: Baseline to Week 13
Population: Phe Responders who are <18 Years of Age
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 29 | 36
T score | -0.7 [-4.0 to 2.7] | -4.8 [-8.0 to -1.6]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.034, ANCOVA; Adjusted for Baseline BRIEF Parent-GEC T Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-7.9 to -0.3], Standard Error of Mean 1.9

7. Secondary Outcome: Change in Attention-Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS) / Adult ADHD Self-Report Scale (ASRS) Total Score From Week 13 to Week 26
Description: Durability of the therapeutic effect of 6R-BH4 on ADHD through 26 weeks in subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  The total ADHD-RS score and the corrected total ARS score range from 0 to 54, with higher scores corresponding to worse severity of ADHD symptoms.
Time Frame: Week 13 to Week 26
Population: Phe Responders with ADHD Symptoms
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm With ADHD Symptoms | Responders in 6R-BH4 20 mg/kg/Day Arm With ADHD Symptoms
Number analyzed (Participants) | 19 | 19
units on a scale | -4.0 [-8.2 to 0.2] | -1.4 [-6.1 to 3.3]
Statistical Analysis 1: Comparison: Responders in Placebo Arm With ADHD Symptoms vs Responders in 6R-BH4 20 mg/kg/Day Arm With ADHD Symptoms; Test type: Superiority or Other; p = 0.312, ANCOVA; Adjusted for Week 13 ADHD RS/ASRS Total Score, age group, and ADHD medication; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-2.6 to 7.8], Standard Error of Mean 2.6

8. Secondary Outcome: Change in Hamilton Anxiety Rating Scale (HAM-A) Score From Week 13 to Week 26
Description: Durability of the therapeutic effect of 6R-BH4 on anxiety through 26 weeks in subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  HAM-A Score is a total score ranging from 0 to 56 with higher scores corresponding to worse severity of anxiety symptoms. The HAM-A has 14 items, each measuring specific anxiety symptom clusters. Each item is given a 5-point-score as: 0, absent; 1, mild; 2, moderate; 3, severe; or 4, incapacitating.
Time Frame: Week 13 to Week 26
Population: Phe Responders
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 60
units on a scale | 0.1 [-1.7 to 1.8] | -0.5 [-2.3 to 1.4]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.590, ANCOVA; Adjusted for Week 13 HAMA Anxiety Rating Scale Total Score, age group, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.4 to 1.4], Standard Error of Mean 1.0

9. Secondary Outcome: Change in Hamilton Depression Rating Scale (HAM-D) Score From Week 13 to Week 26
Description: Durability of the therapeutic effect of 6R-BH4 on depression through 26 weeks in subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  HAM-D Score is a total score ranging from 0 to 48 with higher scores corresponding to worse severity of depression. The HAM-D is a 17-item depression rating scale. Nine of the items are scored on a 5-point scale as: 0, absence of depressive symptom being measured; 1, doubt concerning the presence of the symptom; 2, mild symptoms; 3, moderate symptoms; or 4, severe symptoms. The remaining 8 items are scored on a 3-point scale as: 0, absence; 1, doubt on the presence of the symptom; or 2, clear presence of symptoms.
Time Frame: Week 13 to Week 26
Population: Phe Responders
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 60
units on a scale | 0.1 [-1.3 to 1.5] | 0.5 [-1.1 to 2.0]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.636, ANCOVA; Adjusted for Week 13 HAMD Rating Scale Total Score, age group, ADHD symptom, and ADHD; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.2 to 1.9], Standard Error of Mean 0.8

10. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) From Week 13 to Week 26
Description: Durability of the therapeutic effect of 6R-BH4 on global function through 26 weeks in subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  CGI-S is a 7-point scale that requires the clinician to rate the severity of the subject's mental illness at the time of assessment, relative to clinician's past experience with subjects who have the same diagnosis. Considering total clinical experience, a subject is assessed on the severity of mental illness at the time of rating as: 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 6, severely ill; or 7, among the most extremely ill.
Time Frame: Week 13 to Week 26
Population: Phe Responders
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 60
units on a scale | -0.0 [-0.3 to 0.3] | 0.1 [-0.2 to 0.4]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.510, ANCOVA; Adjusted for Week 13 Global Impression-Severity Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.5], Standard Error of Mean 0.2

11. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF) Adult-Global Executive Composite (GEC) T Score From Week 13 to Week 26
Description: Durability of the therapeutic effect of 6R-BH4 on executive function through 26 weeks in subjects who had a blood Phe level reduction after treatment with 6R-BH4.
  The scoring for the GEC T Score is complex and is achieved using proprietary software designed to generate scores based on raw data collected. Higher scores suggest a higher level of dysfunction.
Time Frame: Week 13 to Week 26
Population: Phe Responders who is >=18 Years of Age
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 28 | 24
T score | -0.7 [-4.5 to 3.1] | 0.9 [-3.7 to 5.4]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.395, ANCOVA; Adjusted for Week 13 BRIEF Adult-GEC T Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-2.1 to 5.2], Standard Error of Mean 1.8

12. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF) Parent-Global Executive Composite (GEC) T Score From Week 13 to Week 26
Description: as for outcome 11
Time Frame: Week 13 to Week 26
Population: Phe Responders who is <18 Years of Age
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 29 | 36
T score | -1.3 [-4.3 to 1.7] | 0.0 [-2.7 to 2.7]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.443, ANCOVA; Adjusted for Week 13 BRIEF Parent-GEC T Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.1 to 4.7], Standard Error of Mean 1.7

13. Secondary Outcome: Change in Attention-Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS) / Adult ADHD Self-Report Scale (ASRS) Total Score From Baseline to Week 26
Description: as for outcome 7
Time Frame: Baseline to Week 26
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm With ADHD Symptoms | Responders in 6R-BH4 20 mg/kg/Day Arm With ADHD Symptoms
Number analyzed (Participants) | 19 | 19
units on a scale | -9.5 [-14.2 to -4.8] | -9.3 [-14.5 to -4.2]
Statistical Analysis 1: Comparison: Responders in Placebo Arm With ADHD Symptoms vs Responders in 6R-BH4 20 mg/kg/Day Arm With ADHD Symptoms; Test type: Superiority or Other; p = 0.953, ANCOVA; Adjusted for Baseline ADHD-RS/ASRS Total Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-5.5 to 5.8], Standard Error of Mean 2.8

14. Secondary Outcome: Change in Hamilton Anxiety Rating Scale (HAM-A) Score From Baseline to Week 26
Description: as for outcome 8
Time Frame: Baseline to Week 26
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 61
units on a scale | -3.9 [-5.8 to -2.0] | -4.2 [-6.3 to -2.2]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.733, ANCOVA; Adjusted for Baseline Hamilton Anxiety Rating Scale (HAM-A) Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.4 to 1.7], Standard Error of Mean 1.0

15. Secondary Outcome: Change in Hamilton Rating Scale For Depression (HAM-D) Score From Baseline to Week 26
Description: as for outcome 9
Time Frame: Baseline to Week 26
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 61
units on a scale | -2.6 [-4.1 to -1.0] | -2.0 [-3.7 to -0.4]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.522, ANCOVA; Adjusted for Baseline Hamilton Rating Scale For Depression (HAM-D) Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.1 to 2.2], Standard Error of Mean 0.8

16. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) From Baseline to Week 26
Description: as for outcome 10
Time Frame: Baseline to Week 26
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 61
units on a scale | -0.6 [-0.9 to -0.3] | -0.5 [-0.8 to -0.2]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.564, ANCOVA; Adjusted for Baseline Clinical Global Impression-Severity (CGI-S), ADHD symptom, and ADHD medication; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.4], Standard Error of Mean 0.2

17. Primary Outcome: Number of Participants With a Score of 1 or 2 in Global Function Evaluation (CGI-I) From Baseline to Week 13.
Description: Effects of 6R-BH4 on global function in PKU subjects in subjects that had a blood Phe level reduction after treatment with 6R-BH4 at screening.
  The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: 13 weeks
Population: Missing data for 1 subject in the Responders in 6R-BH4 20 mg/kg/day Arm
Measure: Number; unit: Number of participants with scale 1 or 2
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 57 | 60
Number of participants with scale 1 or 2 | 15 | 13
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.67, Cochran-Mantel-Haenszel; Adjusted for age group, ADHD symptom, and ADHD medication; Relative Risk = 0.87, 95% CI 2-sided [0.46 to 1.64]

18. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF) Adult-Global Executive Composite (GEC) T Score From Baseline to Week 26
Description: as for outcome 11
Time Frame: Baseline to Week 26
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 28 | 25
T score | -7.1 [-12.6 to -1.6] | -7.7 [-14.5 to -0.9]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.833, ANCOVA; Adjusted for Baseline BRIEF Adult-GEC T Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-6.2 to 5.0], Standard Error of Mean 2.8

19. Secondary Outcome: Change in Behavior Rating Inventory of Executive Function (BRIEF) Parent-Global Executive Composite (GEC) T Score From Baseline to Week 26
Description: as for outcome 11
Time Frame: Baseline to Week 26
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | Responders in Placebo Arm | Responders in 6R-BH4 20 mg/kg/Day Arm
Number analyzed (Participants) | 29 | 36
T score | -2.6 [-6.2 to 1.0] | -4.8 [-8.2 to -1.4]
Statistical Analysis 1: Comparison: Responders in Placebo Arm vs Responders in 6R-BH4 20 mg/kg/Day Arm; Test type: Superiority or Other; p = 0.279, ANCOVA; Adjusted for Baseline BRIEF Parent-GEC T Score, ADHD symptom, and ADHD medication; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-6.3 to 1.8], Standard Error of Mean 2.0

ADVERSE EVENTS:
Time Frame: Study Period
Groups:
- Randomized Treatment Period - Placebo: Randomized Treatment Period - Placebo: Placebo (tablet without active ingredient) is dosed once/day for the first 13 weeks of the study.
- Randomized Treatment Period - 6R-BH4: Randomized Treatment Period - Sapropterin dihydrochloride: A dose of 20 mg/kg/day will be administered. Route of administration is oral (intact).
- Randomized Treatment Period - Overall: Randomized Treatment Period - All patients
- Open-Label Treatment Period - Placebo-6R-BH4: Open-label Treatment Period - Placebo: Placebo (tablet without active ingredient) is dosed once/day for the first 13 weeks of the study.
- Open-Label Treatment Period - 6R-BH4: Open-label Treatment Period - Sapropterin dihydrochloride: A dose of 20 mg/kg/day will be administered. Route of administration is oral (intact).
- Open-Label Treatment Period - Overall: Open-label Treatment Period - All patients
- 6R-BH4 Treatment Period - 6R-BH4: 6R-BH4 Treatment Period - Sapropterin dihydrochloride: A dose of 20 mg/kg/day will be administered. Route of administration is oral (intact).
- 6R-BH4 Treatment Period - Combined: 6R-BH4 Combined Treatments - Sapropterin dihydrochloride: A dose of 20 mg/kg/day will be administered. Route of administration is oral (intact).
Arm/Group | Randomized Treatment Period - Placebo | Randomized Treatment Period - 6R-BH4 | Randomized Treatment Period - Overall | Open-Label Treatment Period - Placebo-6R-BH4 | Open-Label Treatment Period - 6R-BH4 | Open-Label Treatment Period - Overall | 6R-BH4 Treatment Period - 6R-BH4 | 6R-BH4 Treatment Period - Combined
Serious Adverse Events (participants affected / at risk) | 3/108 | 0/98 | 3/206 | 2/104 | 0/95 | 2/199 | 0/98 | 2/202
Other Adverse Events (participants affected / at risk) | 80/108 | 79/98 | 159/206 | 79/104 | 71/95 | 150/199 | 86/98 | 165/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment Period - Placebo (N=108) | Randomized Treatment Period - 6R-BH4 (N=98) | Randomized Treatment Period - Overall (N=206) | Open-Label Treatment Period - Placebo-6R-BH4 (N=104) | Open-Label Treatment Period - 6R-BH4 (N=95) | Open-Label Treatment Period - Overall (N=199) | 6R-BH4 Treatment Period - 6R-BH4 (N=98) | 6R-BH4 Treatment Period - Combined (N=202)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amino acid level increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment Period - Placebo (N=108) | Randomized Treatment Period - 6R-BH4 (N=98) | Randomized Treatment Period - Overall (N=206) | Open-Label Treatment Period - Placebo-6R-BH4 (N=104) | Open-Label Treatment Period - 6R-BH4 (N=95) | Open-Label Treatment Period - Overall (N=199) | 6R-BH4 Treatment Period - 6R-BH4 (N=98) | 6R-BH4 Treatment Period - Combined (N=202)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (5) | 9 (10) | 2 (2) | 7 (7) | 9 (9) | 9 (12) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 10 (12) | 14 (17) | 8 (8) | 4 (6) | 12 (14) | 13 (18) | 21 (26)
Nausea (Gastrointestinal disorders) | 10 (10) | 4 (5) | 14 (15) | 10 (11) | 7 (7) | 17 (18) | 10 (12) | 20 (23)
Vomiting (Gastrointestinal disorders) | 14 (14) | 4 (5) | 18 (19) | 12 (15) | 3 (6) | 15 (21) | 6 (11) | 18 (26)
Pyrexia (General disorders) | 5 (5) | 1 (1) | 6 (6) | 5 (5) | 7 (7) | 12 (12) | 8 (8) | 13 (13)
Nasopharyngitis (Infections and infestations) | 9 (10) | 11 (13) | 20 (23) | 12 (13) | 11 (11) | 23 (24) | 19 (24) | 31 (37)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 4 (5) | 11 (12) | 10 (11) | 3 (4) | 13 (15) | 7 (9) | 17 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 4 (5) | 8 (9) | 6 (7) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 4 (5) | 3 (3) | 7 (9) | 10 (12) | 8 (11) | 11 (14)
Headache (Nervous system disorders) | 28 (37) | 25 (51) | 53 (88) | 16 (21) | 17 (30) | 33 (51) | 32 (81) | 48 (102)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 15 (15) | 8 (8) | 8 (10) | 16 (18) | 10 (17) | 18 (25)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 7 (10) | 18 (22) | 4 (5) | 12 (15) | 16 (20) | 17 (25) | 21 (30)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6) | 16 (16) | 11 (11) | 11 (13) | 22 (24) | 16 (19) | 27 (30)

LIMITATIONS AND CAVEATS:
As specified in the SAP, no multiplicity adjustment was made in the analyses; therefore, the family-wise error rate was not controlled in this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less